CLINICAL TRIAL: NCT04754581
Title: Dynamic in Vivo PET Imaging and ex Vivo Biopsies From Skeletal Muscle and Adipose Tissue to Investigate the Effects of Exercise on Insulin Resistance and Mitochondrial Energetics in Type 2 Diabetes
Acronym: EXPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1581803
Record Dates: First submitted 2021-02-05; First posted 2021-02-15 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise Test; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: This is a single-site, pre-post design pilot study with no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Other)
  Interventions: Other: Maximal ATP Production (ATPmax); Other: Exercise Testing (VO2max); Procedure: Muscle Biopsy; Procedure: Adipose Tissue Biopsy; Other: Hyperinsulinemic euglycemic clamp; Other: PET imaging

INTERVENTIONS:
Other: Maximal ATP Production (ATPmax) — ATPmax will be measured in order to determine in vivo mitochondrial capacity. The magnetic resonance scans to measure mitochondrial energetics will also be performed.
Other: Exercise Testing (VO2max) — Aerobic fitness level will be assessed while participant pedals on a stationary bicycle/walk on a treadmill. The volume of oxygen intake and carbon dioxide (CO2) production will be measured.
Procedure: Muscle Biopsy — Sample muscle cells from the left leg Vastus Lateralis (thigh) muscle.
Procedure: Adipose Tissue Biopsy — Sample fat tissue from the abdomen.
Other: Hyperinsulinemic euglycemic clamp — Measurement of insulin sensitivity.
Other: PET imaging — After an overnight fast, an intravenous catheter will be placed in each arm (one with arterial line for PET infusion, and the other for infusion of insulin, glucose, and 6,6 D2 glucose tracer. FDG-glucose will be injected followed by 90-minute PET scanning of the thigh.

SUMMARY:
The overall aim of this pilot study is to investigate the effects of exercise training on skeletal muscle and adipose tissue insulin resistance in subjects with Type 2 Diabetes (T2D).

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-65 years
2. Men and women
3. Body mass index (BMI) between 25 and 45 kg/m2
4. Sedentary (1 day or less per week of structured exercise)
5. Type 2 diabetes mellitus determined by self-report or by a fasting glucose >126mg/dl
6. Weight stable (± 2 kg) for prior 3 months
7. Willing to commit to the schedule of assessment visits, including the exercise intervention

Exclusion Criteria:

1. Currently taking insulin, injectable incretin mimetics and thiazolidinediones
2. Taking more than two glucose-lowering medications
3. Resting blood pressure ≥ 160/100 mm Hg
4. Triglycerides ≥ 500 mg/dL
5. Any renal, cardiac, liver, lung, or neurological disease that in the opinion of the principal investigator would compromise participant safety or the participants' ability to complete the exercise training protocol
6. Any significant disease or unstable medical condition (i.e., coronary heart disease, chronic renal failure, chronic hepatic disease, severe pulmonary disease)
7. Presence of clinically significant abnormalities on electrocardiogram (ECG) that is a contra-indication to exercise training
8. Pulse check ("Allen test") indicates participant has poor blood flow in the hands
9. Cancer (active malignancy with or without concurrent chemotherapy; except for basal cell carcinoma)
10. Pregnancy during the previous 6 months, lactating, or planned pregnancy in the next year
11. Use of drugs known to affect energy metabolism or body weight: including, but not limited to orlistat, sibutramine, ephedrine, phenylpropanolamine, corticosterone, etc
12. Current treatment with blood thinners or anti-platelet medications that cannot be safely stopped for testing procedures
13. Participant is currently taking anti-inflammatory medication or has had inflammatory medication within 1 week prior to screening (including over the counter formulations: e.g. Aleve, Motrin, Ibuprofen, Naproxen, low dose ASA.
14. New onset (<3 months on a stable regime) hormone replacement therapy
15. Current use of beta-adrenergic blocking agents
16. Major surgery on the abdomen, pelvis, or lower extremities within previous 3 months
17. Increased liver function tests (AST/ALT/GGT/or alkaline phosphatase greater than 2.5 times the upper limit of normal)
18. Abnormal blood count/anemia, blood transfusion or blood donation within the last 2 months
19. Current smokers (smoking within the past 3 months prior to screening visit, including any/all tobacco products)
20. Current drug or alcohol abuse/dependence
21. Metal implants (pace-maker, aneurysm clips) based on investigator's judgment at screening
22. Not physically capable of performing the exercise required of the study protocols
23. Plans to be away >2 weeks in the next 3 months
24. Unable to participate in Magnetic Resonance Imaging (MRI) assessments due to physical limitations of equipment tolerances (e.g. MRI bore size) based on investigator's judgment at screening.
25. Unable to tolerate MRI or claustrophobia.
26. Nickel allergy
27. Lidocaine allergy
28. Unable or unwilling to communicate with staff or to provide written informed consent

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Individual steps of muscle glucose uptake (pre-exercise) | 24 hours
  Muscle glucose uptake will be assessed two times (pre and post exercise intervention) on the biceps femoris and vastus lateralis through PET imaging and hyperinsulinemic euglycemic clamp.
Individual steps of muscle glucose uptake (post-exercise) | 24 hours
  Muscle glucose uptake will be assessed two times (pre and post exercise intervention) on the biceps femoris and vastus lateralis through PET imaging and hyperinsulinemic euglycemic clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Bret Goodpaster, PhD, Principal Investigator — Scientific Director | Senior Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

REFERENCES:
- See also: Website for AdventHealth Translational Research Institute — https://www.adventhealthresearchinstitute.com/research/translational-research